CLINICAL TRIAL: NCT05590533
Title: Validity and Reliability of the Turkish Version of F-2-MS Scale
Brief Title: Turkish Version of F-2-MS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, Assoc. Prof., Pamukkale University
Other Study IDs: 19.10.2022/F-2-MS
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Cultural Adaptation; Reliability; Validity; Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cultural adaptation, reliability and validity — Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of the F-2-MS

SUMMARY:
The aims of this study were to perform cultural adaptation of the F-2-MS and provide information regarding the factor structure, reliability and validity of the instrument in Turkish speaking patients with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 20-65 years, with an EDSS score of 0-5, who have not had an attack in the last 2 months, who have no cognitive problems (a score of 6 or more according to the Hodkinson Mental Test), who do not have additional neurological diseases other than MS, and who volunteer to participate in the study will be included.

Exclusion Criteria:

* Individuals with an EDSS score greater than 5, who are in the attack period, who have vestibulosupressant or drug or alcohol use habits that cause neuropathy, and who have communication problems will be excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with multiple sclerosis with an EDSS score of 5 or less
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
F-2-MS Scale | 10 minutes
  F-2-MS is a novel scale to assess fatigue and perceived fatigability in patients with MS

IPD SHARING:
Plan to Share IPD: No